CLINICAL TRIAL: NCT05875974
Title: A Prospective, Open-Label, Single-Arm, Multicenter Study to Evaluate the Effect of Low-Sodium Oxybate Oral Solution (XYWAV) on Sleepiness, Polysomnography, and Functional Outcomes in Adult Participants Aged 18 to 75 Years With Idiopathic Hypersomnia or Narcolepsy
Brief Title: A Study to Investigate the Effect of XYWAV on Sleepiness, Polysomnography, and Functional Outcomes in Participants With Idiopathic Hypersomnia or Narcolepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JZP258-407
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Hypersomnia; Narcolepsy
Keywords: Idiopathic Hypersomnia; Narcolepsy; Excessive daytime sleepiness; Polysomnography; JZP258; XYWAV; Oxybate
MeSH Terms: conditions — Idiopathic Hypersomnia; Narcolepsy; Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JZP258 (Experimental): Participants will self-administer an oral dose of JZP258 (XYWAV) as per label and titrate to an optimal dosage for each participant.
  Interventions: Drug: JZP258 (XYWAV)

INTERVENTIONS:
Drug: JZP258 (XYWAV) — Narcolepsy Cohort: Initiate dosage per XYWAV label and titrate to effect.
  IH Cohort: Initiate dosage per XYWAV label and titrate to effect.
  Narcolepsy >9-Gram Cohort: XYWAV titrated to a dosage of >9 to 12 grams.

SUMMARY:
This study will assess the safety and efficacy of JZP258 (XYWAV) on sleepiness, polysomnography, and functional outcomes in patients with idiopathic hypersomnia (IH) or narcolepsy.

DETAILED DESCRIPTION:
This prospective, multicenter, single-arm, open-label interventional study will assess the safety and efficacy of JZP258 on sleepiness, polysomnography measurements (eg, sleep stage transitions, sleep patterns, and sleep quality), daytime and nighttime symptoms, pharmacokinetics (in narcolepsy), and patient-reported outcomes that include subjective sleep quality and quality of life in patients with IH or narcolepsy.

ELIGIBILITY:
Key Inclusion Criteria:

* Is 18 to 75 years of age (inclusive) at the time of signing the informed consent form (ICF)
* Has a primary diagnosis of IH meeting International Classification of Sleep Disorders, Third Edition (ICSD-3) criteria or narcolepsy (Type 1 or Type 2) meeting ICSD-3 or Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria.
* If not currently taking oxybate medication, has clinically significant symptoms of Excessive daytime sleepiness (EDS) with an ESS score > 10 at Screening Visit 1. If currently taking oxybate medication, has an ESS score > 10 at the Baseline Visit 2 polysomnography (after washout period). Note: Not applicable for participants entering the Narcolepsy >9-gram cohort (see additional criteria below for the Narcolepsy >9-gram cohort).
* If currently treated with anticataplectics and/or alerting agents, has been taking the same dosage for at least 1 month prior to Screening Visit 1 and has no current plans to adjust the dosage during the study period. Note: Alerting agents refer to either traditional stimulants (eg, amphetamines, methylphenidates) or wake-promoting agents (eg, modafinil, pitolisant, solriamfetol).

Additional Inclusion Criteria for Participants in the Narcolepsy >9-Gram Cohort

* Is on a current treatment regimen including XYWAV at a dosage of 9 grams

Key Exclusion Criteria:

* Shows evidence of a previous untreated or inadequately treated sleep disorder considered by the investigator to negatively impact the conduct of the study, including sleep-disordered breathing, parasomnias, circadian rhythm sleep disorders, or restless legs syndrome determined by a previous sleep-laboratory diagnosis or interview utilizing modules of the Diagnostic Interview for Sleep Patterns and Disorders.
* Shows evidence of untreated or inadequately treated sleep-disordered breathing during Baseline Visit 2 polysomnography defined as an Apnea/Hypopnea Index (AHI) > 10, using the US Centers for Medicare and Medicaid Services rules (CMS.gov).
* Has a history or presence of any unstable or clinically significant medical condition (chronic pain condition that may impact sleep), behavioral or psychiatric disorder (including active suicidal ideation or current or past [within 1 year] major depressive episode), or history or presence of another neurologic disorder or surgical history that might affect the participant's safety and/or interfere with the conduct of the study, in the opinion of the investigator.
* Has recently taken (ie, within 1 month prior to screening), is taking, or plans to take any of the following:

  * A substance or medication contraindicated with XYWAV use, ie. specifically alcohol and sedative hypnotics
  * A medication with a known drug-drug interaction with XYWAV
  * A medication that may have similar EEG effects to XYWAV
  * Medications known to have clinically significant CNS sedative effects
  * Other medications, natural health products, or substances from which the participant experiences clinically significant sedation

Additional Exclusion Criterion for Participants in the Narcolepsy >9-Gram Cohort

• Any past or current medical conditions or experience that, in the investigator's clinical judgment, would preclude further increases in the current oxybate medication dosage beyond 9 grams

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale (ESS) Total Score in Participants With IH and Narcolepsy Treated With XYWAV | Baseline up to End of Treatment (approximately 10-36 weeks)

SECONDARY OUTCOMES:
Idiopathic Hypersomnia Severity Scale (IHSS) Total Score in Participants With IH Treated With XYWAV | Baseline up to End of Treatment (approximately 10-21 weeks)
Number of Stage Shifts of Sleep in Participants With Narcolepsy Treated With XYWAV | Baseline up to End of Treatment (approximately 10-36 weeks)
Duration of Sleep Stages in Participants With Narcolepsy Treated With XYWAV | Baseline up to End of Treatment (approximately 10-36 weeks)
Number of Nocturnal Awakenings and Nocturnal Arousals in Participants With Narcolepsy Treated With XYWAV | Baseline up to End of Treatment (approximately 10-36 weeks)
Percentage of Sleep Stages in Participants With Narcolepsy Treated With XYWAV | Baseline up to End of Treatment (approximately 10-36 weeks)
Patient Global Impression of Change (PGI-C) Score in Participants With IH and Narcolepsy Treated With XYWAV (Overall, Sleep Inertia, and Fatigue) | End of Treatment (approximately 10-36 weeks)
Level of Rested or Refreshed Upon Awakening in Participants With IH and Narcolepsy Treated With XYWAV (Sleep Diary) | Baseline up to End of Treatment (approximately 10-36 weeks)
Patient Global Impression of Severity (PGI-S) Score in Participants With IH and Narcolepsy Treated With XYWAV (Overall, Sleep Inertia, and Fatigue) | Baseline up to End of Treatment (approximately 10-36 weeks)
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) In a Subset of Participants With Narcolepsy Treated With XYWAV | PK: Predose, 0.5 hour, 0.75 hour, 1 hour, 1.5 hour post-first dose and post-second dose, 6 hour post-first dose, 8 hour post-first dose
Pharmacokinetic Parameter Area Under the Concentration-Time Curve From time 0 to Infinity (AUC0-inf) In a Subset of Participants With Narcolepsy Treated With XYWAV | PK: Predose, 0.5 hour, 0.75 hour, 1 hour, 1.5 hour post-first dose and post-second dose, 6 hour post-first dose, 8 hour post-first dose

CONTACTS AND LOCATIONS:
Locations (32):
- United States (29):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Perseverance Research Center, LLC, Scottsdale, Arizona
  - Amnova Clinical Research, Irvine, California
  - Long Beach Research Institute, Lakewood, California
  - Santa Monica Clinical Trials, Los Angeles, California
  - Stanford School of Medicine, Redwood City, California
  - TriValley Sleep Center, San Ramon, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Meris Clinical Research, LLC, Brandon, Florida
  - PharmaDev Clinical Research Institute, LLC, Miami, Florida
  - Florida Hospital for Children, Winter Park, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Centricity Research Rincon - DBA IACT Health Southeast Lung Associates Research, Rincon, Georgia
  - Neurocare, Inc., dba Neurocare Center for Research, Newtown, Massachusetts
  - Clinical Neurophysiology Services, P.C., Sterling Heights, Michigan
  - St. Lukes Hospital Medical Center, Chesterfield, Missouri
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Stern Research Partners, LLC, Huntersville, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - Cleveland Clinic Main Campus - Clinical Research Unit, Cleveland, Ohio
  - Ohio Sleep Medicine and Neuroscience Institute, Dublin, Ohio
  - Abington Neurological Associates, LTD, Abington, Pennsylvania
  - Geisinger Clinic, Scranton, Pennsylvania
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Comprehensive Sleep Medicine Associates, Houston, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Tricoastal Narcolepsy and Sleep Disorders Center, Sugar Land, Texas
- Canada (3):
  - Heritage Medical Research Clinic, University of Calgary, Calgary, Alberta
  - AMNDX Inc, Markham, Ontario
  - Johda Tishon Inc, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No